CLINICAL TRIAL: NCT07052500
Title: Investigating the Impact of Seed Cycling on Menstrual Regularity, Dysmenorrhea, and Premenstrual Symptoms
Brief Title: Impact of Seed Cycling on Menstrual Regularity, Dysmenorrhea, and Premenstrual Symptoms
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Loma Linda University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 5250289
Record Dates: First submitted 2025-06-26; First posted 2025-07-04 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Menstruation Disorders; Menstrual Cramps; Menstruation
Keywords: Seed Cycling; Menstrual Regularity; Dysmenorrhea; Premenstrual Symptoms
MeSH Terms: conditions — Menstruation Disturbances; Dysmenorrhea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Seed Cycling single arm intervention (Experimental): Subjects will receive sunflower seeds, pumpkin seeds, flaxseed and sesame seeds during the intervention
  Interventions: Dietary Supplement: Seed Cycling

INTERVENTIONS:
Dietary Supplement: Seed Cycling — Daily consumption of 1 tablespoon each of flax and pumpkin seeds during the follicular phase and 1 tablespoon each of sunflower and sesame seeds during the luteal phase

SUMMARY:
The purpose of this research is to investigate the impact of seed cycling on menstrual regularity, cramps, and pre-menstrual symptoms in women with an irregular menstrual cycle and/or dysmenorrhea. The research seeks to provide evidence-based insights into the potential benefits of seed cycling as a holistic approach to women's reproductive health.

It is expected that your participation will last 3 months. Procedures and Activities. You will be provided with and asked to consume specific seeds daily. The seeds are to be consumed as follows: follicular phase (the period from the first day of menstruation (day 1) to ovulation (day 14) in a typical 28-day cycle): 1 tablespoon flax seeds and 1 tablespoon pumpkin seeds, and luteal phase (the period between ovulation and the start of the next period; typically days 15-28): 1 tablespoon sunflower seeds and 1 tablespoon sesame seeds. Before the intervention and once monthly for a total of 3 cycles, you will be asked to complete an online menstrual health symptom questionnaire (MHSQ) and keep track of your menstrual cycle days on the built-in health tracking app on your electronic device.

Risks. Some of the foreseeable risks or discomforts of your participation include the potential for mild gastrointestinal side effects, the potential for allergic reactions, and the possibility of no significant benefit.

Benefits. Possible benefits include the potential for improved menstrual cycle regularity, the potential for a reduction in premenstrual syndrome (PMS) symptoms, and the potential for nutritional benefits. Societal benefits include additional knowledge on seed cycling to help manage menstrual regularity and PMS symptoms.

DETAILED DESCRIPTION:
This study will employ a single-arm intervention design. As a single-arm study, all enrolled participants will receive the same seed cycling intervention, and there will be no separate control or comparison group. Data collection will occur over three menstrual cycles for each participant, starting from their individual cycle start dates.

The study duration is approximately three months from September 2025 to December 2025. Data collection will involve a combination of:

• Pre- and Post-Intervention Surveys: Participants will complete a Menstrual Health Symptom Questionnaire (MHSQ)8 via Google Forms. The pre-survey will be administered prior to the intervention, and cycle-end surveys will be conducted at 1-month, 2-month, and 3-month follow-ups after starting the seed cycling intervention.

• Monthly Tracking: Participants will utilize the built-in health tracking app on their electronic device to track their cycle days on the menstrual cycle tracking feature. This tool will facilitate the tracking of period cycle days and will also be used for ongoing tracking of symptoms, supplementing the monthly survey data.

• Individual Email Reminders: To enhance compliance and data completeness, individual email reminders will be sent to participants on a biweekly basis.

e. Study Procedures and Schedule This study involves a series of structured visits and ongoing self-monitoring to assess the impact of the seed cycling intervention on menstrual cycle regularity and associated symptoms. All procedures related to the seed cycling intervention and associated data collection are considered experimental and specifically designed for the purpose of this research study. There are no elements of "routine care" integrated into this study, as the intervention itself is not a standard medical practice.

Measures and Timeframes

The following specific tests and measures will be carried out:

•

Menstrual Health Symptom Questionnaire (MHSQ):

This is a validated, self-administered questionnaire administered online via Google Forms. It collects detailed information on participants' menstrual cycle regularity, duration, associated symptoms (e.g., lower abdomen pain, breast tenderness, muscle pain, nausea, bone pain, feeling bloated, diarrhea, joint pain, headaches, constipation, feeling excessively sad, feeling emotionally unstable, feeling irritable or short-tempered, feeling anxious, being excessively hungry or feeling lack of hunger, having insomnia, and feeling excessively tired) and their severity.

▪

Timeframes:

• Baseline/Pre-intervention: Completed at Visit 1 (Day 1). This MHSQ will serve as the baseline measure for all menstrual health symptoms and cycle characteristics.

• Post-intervention/Follow-up: Completed at Visit 2 (Day 28), Visit 3 (Day 56), and at the End of Study (Day 84 or last day of the third cycle).

• Acceptable Window: Completion of the MHSQ is expected on the scheduled day of each visit. A window of ± 2 days from the scheduled day for online completion is considered acceptable to account for unforeseen participant availability, but efforts will be made to ensure timely completion.

•

Menstrual Cycle Tracking via smartphone health tracking app:

▪ Menstrual Cycle Days: Start and end dates of menstruation.

▪ Symptom Tracking: Daily or periodic recording of menstrual symptoms as outlined in the MHSQ (serving as a supplementary, continuous record to the periodic MHSQ completions).

▪

Timeframes:

• Orientation and study overview for participants will occur on Visit 1 (Day 1) in the Nichol Hall Kitchen. Participants will be instructed to begin tracking immediately after training.

• Throughout the Study: Participants will continuously track their cycles and symptoms from Day 1 until the end of study (Day 84 or last day of the third cycle).

• Verification: At Visit 2 (Day 28) in the Nichol Hall Kitchen, accuracy of use of the menstrual cycle tracking feature on the participants' smartphone health tracking apps will be verified. This will allow for real-time feedback and correction if tracking issues are identified.

▪ Acceptable Window: Daily tracking is expected. Minor gaps of 1-2 days in tracking may be acceptable if clear recall allows for accurate back-entry, but consistent daily logging will be encouraged.

Experimental Procedures

All components of the intervention and data collection are experimental procedures for the purpose of this study:

Provision of Seed Cycling Intervention Materials:

▪

Timeframes:

• Visit 1 (Day 1): Provision of 1 month (28 days) of individually packaged and labeled seeds with the corresponding seed cycling schedule.

• Visit 2 (Day 28): Provision of the second month's supply of seeds (28 days) and schedule. If the menstrual cycle has not started by day 28, additional sunflower and sesame seeds will be provided for use until the next cycle commences.

• Visit 3 (Day 56): Provision of the third month's supply of seeds (28 days) and schedule. If the menstrual cycle has not started by day 56, additional sunflower and sesame seeds will be provided for use until the next cycle commences.

▪ This involves the distribution of specific, pre-portioned seeds (flax, pumpkin, sesame, and sunflower) according to the predefined seed cycling schedule. The packaging and labeling will ensure adherence to the correct sequence and dosage.

ELIGIBILITY:
Inclusion Criteria:

* Women ages 18-45 with an irregular menstrual cycle and/or menstrual cramps, and/or pre-menstrual symptoms. "Irregular"is defined as a cycle that deviates from the typical pattern of 21 to 35 days between periods
* Access to an electronic device with a built-in health tracking app that can connect to the internet and is capable of reading QR codes
* Speak and understandEnglish

Exclusion Criteria:

* Current or recent use (within the last 3 months) of hormonal birth control or hormone replacement therapy
* Currently pregnant, lactating, or planning pregnancy between now and December 2025
* Active gastrointestinal (GI) condition
* Currently consuming seed oil supplements
* Allergic to flax seeds, pumpkin seeds, sesame seeds, or sunflower seeds
* Unable to chew or swallow flax seeds, pumpkin seeds, sesame seeds, or sunflower seeds
* Daily, regular consumption of flax seeds, pumpkin seeds, sesame seeds, or sunflower seeds

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-05 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Change in menstrual cycle from irregular to regular | 3 months
  The primary endpoint for this study is the proportion of participants reporting a shift to regular menstrual cycles (defined as 21-35 days) after the 3-cycle intervention. This endpoint directly measures the efficacy of the intervention in achieving the primary objective: to determine the proportion of women who self-report a change from irregular to predominantly regular cycles.

SECONDARY OUTCOMES:
Change in menstrual cramp severity | 3 months
  Change in menstrual cramp severity will be assessed using a validated pain scale administered during menstruation, comparing severity during the intervention cycles to the participants' self-reported historical experience. This Page 4 of 16 endpoint will evaluate the intervention's impact on a key symptom associated with menstrual cycles.
Change in pre-menstrual symptoms | 3 months
  Change in pre-menstrual symptoms including lower abdomen pain, breast tenderness, muscle pain, nausea, bone pain, feeling bloated, diarrhea, joint pain, headaches, constipation, feeling excessively sad, feeling emotionally unstable, feeling irritable or short-tempered, feeling anxious, being excessively hungry or feeling lack of hunger, having insomnia, and feeling excessively tired. Participants will report on the presence and severity of these symptoms using a standardized questionnaire. This endpoint will assess the broader influence of the intervention on overall well-being before and during the menstrual cycle.

CONTACTS AND LOCATIONS:
Locations (1):
- School of Allied Health Professions, Loma Linda, California, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared due to concerns about participant privacy, potential for re-identification, and the risk of data misuse.

REFERENCES:
- [Background] Cassioli E, Rossi E, Melani G, Faldi M, Rellini AH, Wyatt RB, Oester C, Vannuccini S, Petraglia F, Ricca V, Castellini G. The menstrual distress questionnaire (MEDI-Q): reliability and validity of the English version. Gynecol Endocrinol. 2023 Jun 19;39(1):2227275. doi: 10.1080/09513590.2023.2227275. PMID 37356456
- [Background] Itani R, Soubra L, Karout S, Rahme D, Karout L, Khojah HMJ. Primary Dysmenorrhea: Pathophysiology, Diagnosis, and Treatment Updates. Korean J Fam Med. 2022 Mar;43(2):101-108. doi: 10.4082/kjfm.21.0103. Epub 2022 Mar 17. PMID 35320895
- [Background] Attia GM, Alharbi OA, Aljohani RM. The Impact of Irregular Menstruation on Health: A Review of the Literature. Cureus. 2023 Nov 20;15(11):e49146. doi: 10.7759/cureus.49146. eCollection 2023 Nov. PMID 38130524
- [Background] Vaziri F, Zamani Lari M, Samsami Dehaghani A, Salehi M, Sadeghpour H, Akbarzadeh M, Zare N. Comparing the effects of dietary flaxseed and omega-3 Fatty acids supplement on cyclical mastalgia in Iranian women: a randomized clinical trial. Int J Family Med. 2014;2014:174532. doi: 10.1155/2014/174532. Epub 2014 Aug 13. PMID 25197571
- [Background] Matar SS, Farrag AA, Hafez SM, Fahmy RM. The Bioactive Effect of Flaxseed on Women with the Polycystic Ovarian Syndrome. Egyptian Journal of Nutrition. 2021;36(3):49-77. doi: 10.21608/enj.2021.209919
- [Background] Haidari F, Banaei-Jahromi N, Zakerkish M, Ahmadi K. The effects of flaxseed supplementation on metabolic status in women with polycystic ovary syndrome: a randomized open-labeled controlled clinical trial. Nutr J. 2020 Jan 24;19(1):8. doi: 10.1186/s12937-020-0524-5. PMID 31980022
- [Background] Phipps WR, Martini MC, Lampe JW, Slavin JL, Kurzer MS. Effect of flax seed ingestion on the menstrual cycle. J Clin Endocrinol Metab. 1993 Nov;77(5):1215-9. doi: 10.1210/jcem.77.5.8077314.
- [Background] Rasheed N, Ahmed A, Nosheen F, Imran A, Islam F, Noreen R, Chauhan A, Shah MA, Amer Ali Y. Effectiveness of combined seeds (pumpkin, sunflower, sesame, flaxseed): As adjacent therapy to treat polycystic ovary syndrome in females. Food Sci Nutr. 2023 Mar 25;11(6):3385-3393. doi: 10.1002/fsn3.3328. eCollection 2023 Jun. PMID 37324929